CLINICAL TRIAL: NCT04617756
Title: Safety & Efficacy of Neoadjuvant Immunotherapy With Durvalumab (MEDI 4736) Combined With Neoadjuvant Chemotherapy (Gemcitabine/Cisplatin or Gemcitabine/Carboplatin) in Patients With Operable, High-risk, Localized Urothelial Carcinoma of the Upper Urinary Tract
Brief Title: Safety & Efficacy of Durvalumab+Neoadjuvant Chemotherapy for High-risk Urothelial Carcinoma of the Upper Urinary Tract
Acronym: iNDUCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other); Bichat Hospital (Other); Hopital Foch 92151 Suresnes (Unknown); Institut Paoli-Calmettes (Other); European Georges Pompidou Hospital (Other); Saint-Louis Hospital, Paris, France (Other); Centre Hospitalier Lyon Sud (Other); Center Eugene Marquis (Other); IUCT ONCOPOLE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIVI/2018/NH-1
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Urothelial Carcinoma; Cancer
Keywords: Durvalumab; Gemcitabine; Cisplatin; Chemotherapy
MeSH Terms: conditions — Carcinoma, Transitional Cell; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with an estimated glomerular filtration rate equal to or over 60 ml/min./1.73² (cohort 1) will receive treatment combining Durvalumab and gemcitabine with Cisplatin.
  Patients with an estimated glomerular filtration rate of under 60 ml/min./1.73² and over 40 ml/min./1.73² (cohort 2) will receive treatment combining Durvalumab and gemcitabine with Carboplatin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Durvalumab+Gemcitabine/Cisplatin or with Gemcitabine/Carboplatin (Experimental): This is a single arm including 2 different cohorts : Cohort 1 includes patients on 40mg/ML Gemcitabine/50mg Cisplatin used in combination with 50 mg/mL of intravenous Durvalumab (laboratory code MEDI 4736) every 3 weeks for a total of 4 cycles and Cohort 2 includes patients on 40mg/ML Gemcitabine/450mg Carboplatin used in combination with 50 mg/mL of intravenous Durvalumab (laboratory code MEDI 4736) every 3 weeks for a total of 4 cycles..
  Interventions: Drug: Patients receiving neoadjuvant therapy before radical nephrectomy

INTERVENTIONS:
Drug: Patients receiving neoadjuvant therapy before radical nephrectomy — Chemotherapy using either a combination of Gemcitabine/Cisplatin and neoadjuvant immunotherapy therapy with Durvalumab (MEDI 4736) or Chemotherapy with either Gemcitibine/Carboplatin and neoadjuvant immunotherapy therapy with Durvalumab (MEDI 4736)

SUMMARY:
Following radical nephrectomy (RNU) for upper tract urothelial carcinoma (UTUC) most patients face a poor prognosis. Indeed, patients who have undergone RNU for UTUC have 5-year recurrence-free and cancer specific survival probabilities of 69% and 73% respectively.

The primary objective of this study is to assess the pathological complete response rate to combination therapy with neoadjuvant durvalumab and chemotherapy (Gemcitabine/Cisplatin) before surgery in patients with high-risk, localized, non-metastatic urothelial carcinomas of the upper tract.

DETAILED DESCRIPTION:
Following radical nephrectomy (RNU) for upper tract urothelial carcinoma (UTUC) most patients face a poor prognosis. Indeed, patients who have undergone RNU for UTUC have 5-year recurrence-free and cancer specific survival probabilities of 69% and 73% respectively. Additional systemic therapy therefore seems justified for prolonged cancer control. However, there have been very few studies on neoadjuvant/adjuvant therapies in UTUC. Recently, the UK's multicentric POUT trial reported the benefits of adjuvant chemotherapy in UTUC patients. Level 1 evidence has been provided for neoadjuvant therapy for urothelial carcinoma of the bladder via meta-analysis in 2005 but there are also several arguments for systemic therapy in this context especially as most patients lose the function of one kidney and cannot receive nephrotoxic cisplatin-based chemotherapy. Urothelial carcinoma of the upper tract have a different genetic background from carcinomas of the lower tract. The investigators hypothesized that there would be a greater occurrence of lower pathological stages among study group patients who receive neoadjuvant combined Durvalumab/Gemcitabine/Cisplatin or Carboplatin prior to RNU compared to the current literature (Gregg et al. 2018, Almassi et al. 2018). The primary objective is to assess the pathological complete response rate (ypT0) in each cohort and independently of a combination therapy with neoadjuvant durvalumab and chemotherapy (Gemcitabine/Cisplatin) before surgery in patients with high-risk, localized, non-metastatic urothelial carcinomas of the upper tract.Secondary objectives include: assessing partial response rate to treatment, assessing the safety and tolerability of the treatment and evaluating the overall survival, bladder recurrence and dissemination at two years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been correctly informed and has given signed consent.
* Patient is covered by a health insurance scheme.
* Patients aged over 70 must have a G8 score (Soubeyran et al. 2014) of at least 14.
* Patient's body weight must be over 30kg
* Patient has high-grade urothelial carcinoma of the renal pelvis or ureter confirmed histologically (uteroscopic biopsy) or cytologically (urine cytology).
* Presence of divergent histologies (i.e. squamous cell tumour, adenocarcinoma, small cell carcinoma, micropapillary variant) may also give rise to inclusion if there is a high prevalence (over 90%) of a urothelial component.
* Presence of EITHER high-grade disease on the uteroscopic tumor biopsy
* OR Presence of high-grade disease on urine cytology AND infiltrative aspect of renal pelvis/ ureteral wall on the CT scan (presence of hydronephrosis will be considered invasive by definition) with negative cystoscopy.
* Or in the absence of histological evidence, the opinion of the multidisciplinary consultation meeting (RCP) will prevail for the analysis of the imaging and the potential inclusion of the patient in the study
* No prior systemic therapies.
* ECOG performance status 0 to 1.
* M0 No or N1 disease on CT scan.

  * Required initial laboratory values :
* Absolute neutrophil count of over 1500 cells/mm²
* Platelet count of over 100,000 cells/mm3
* Hemoglobin over 9.0 g/dL
* Bilirubin below 1.5 times the Upper Limit of Normal for the institution
* Aspartase transaminase (ASAT) and Alanine transaminase (ALAT) below 2.5 x the Upper Limit of Normal for the institution.
* Alkaline phosphatase below 2.5 times the Upper Limit of Normal for the institution
* INR and aPTT below 1.5 times the Upper Limit of Normal for the institution.
* For Cohort 1 : An estimated glomerular filtration rate of over 60ml/min/1.73m² using the CKD-EPI and/or MDRD equation.
* For Cohort 2 : An estimated glomerular filtration rate of 40ml to 60ml/min/1.73m² using the CKD-EPI and/or MDRD equation.
* Patients with reproductive potential must use an effective method to avoid pregnancy for the duration of the trial.
* Patients must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

* The patient is participating in another interventional trial;
* or is in an exclusion period determined by a previous study;
* or is under judicial protection, or is an adult under guardianship
* or refuses to sign the consent;
* or it is impossible to correctly inform the patient.
* The patient is pregnant or breastfeeding.
* Concomitant diagnosis of muscle invasive or in situ or high grade non muscle invasive urothelial carcinoma of the bladder.
* Evidence of NYHA functional class III or IV heart disease.
* Serious intercurrent medical or psychiatric illness, including serious active infection.
* Concomitant use of any other investigational drugs.
* Diagnosis of immunodeficiency or received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Additional malignancy within last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ cervical cancer that has undergone potentially curative therapy, stable (as defined by PSA change, checked within 30 days) and untreated very low-risk or low-risk prostate cancer defined by current NCCN guidelines. Previous or concomitant history of non-muscle invasive bladder cancer is acceptable.
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception. Subjects that require systemic corticosteroids at physiologic doses not exceed 10mg/day of prednisone or its equivalent would not be excluded from the study. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C.
* Live vaccine received within 30 days prior to the first dose of trial treatment.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of treatment. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Uncontrolled intercurrent illness, including but not limited to, on-going or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response in Cohort 1 | Week 14 - 18
  For Cohort 1 (patients on treatment combining Durvalumab and Gemcitabine associated with Cisplatin) the rate of patients with pathological complete response will be calculated and presented with associated 95% confidence interval on the subpopulation of patients with ureteroscopic biopsy at diagnosis.Pathological complete response is defined as no residual signs of viable tumor cells in tissue samples removed during surgery after treatment. To find out if there is a pathologic complete response, a pathologist will perform an evaluation of the tissue samples under a microscope to see if there are still cancer cells left after the treatment.
Pathological complete response in Cohort 2 | Week 14 - 18
  For Cohort 2 (patients on treatment combining Durvalumab and Gemcitabine associated with Carboplatin) the rate of patients with pathological complete response will be calculated and presented with associated 95% confidence interval on the subpopulation of patients with ureteroscopic biopsy at diagnosis.Pathological complete response is defined as no residual signs of viable tumor cells in tissue samples removed during surgery after treatment. To find out if there is a pathologic complete response, a pathologist will perform an evaluation of the tissue samples under a microscope to see if there are still cancer cells left after the treatment.

SECONDARY OUTCOMES:
Partial pathological response in Cohort 1 | Week 3
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Partial pathological response in Cohort 2 | Week 3
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Partial pathological response in Cohort 1 | Week 6
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Partial pathological response in Cohort 2 | Week 6
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Partial pathological response in Cohort 1 | Week 9
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Partial pathological response in Cohort 2 | Week 9
  Pathological partial response is defined as downstaging to neoadjuvant pathologic stage groups ≤ ypT1N0M0 (ypT0-Ta-Tis/T1 disease).The rate of patients with partial pathological response will be calculated on the subpopulation of patients with ureteroscopic biopsy at diagnosis.
Safety and tolerability of treatment - Cohort 1 | Week 3
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Safety and tolerability of treatment - Cohort 2 | Week 3
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Safety and tolerability of treatment - Cohort 1 | Week 6
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Safety and tolerability of treatment - Cohort 2 | Week 6
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Safety and tolerability of treatment - Cohort 1 | Week 9
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Safety and tolerability of treatment - Cohort 2 | Week 9
  The safety and tolerability of treatment will be assessed by analysing and interpreting Common Terminology Criteria for Adverse Event (CTCAE) until surgery using the National Cancer Institute, Division of Cancer Treatment and Diagnosis (DCTD) listing of CTCAE (NCI CTCAE V5.0).
Treatment success - Overall Survival in Cohort 1 | 2 years after surgery.
  The overall Survival rate of Cohort 1 patients will be collected.
Treatment success - bladder recurrence and dissemination in Cohort 1 | 2 years after surgery.
  Bladder recurrence and dissemination in Cohort 1 patients will be collected.
Treatment success - Overall Survival in Cohort 2 | 2 years after surgery.
  The overall Survival rate of Cohort 2 patients will be collected.
Treatment success - bladder recurrence and dissemination in Cohort 2 | 2 years after surgery.
  Bladder recurrence and dissemination will be collected.
Intercycle report : Blood cells & Platelets in Cohort 1 | Week 3
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report : Blood cells & Platelets in Cohort 2 | Week 3
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report : Electrolytes in Cohort 1 | Week 3
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report : Electrolytes in Cohort 2 | Week 3
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report : Liver in Cohort 1 - AST | Week 3
  - Hepatic workup: Aspartate Aminotransferase (AST) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - ALT | Week 3
  - Hepatic workup: Alanine Aminotransferase (ALT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 -GGT | Week 3
  - Hepatic workup: Gamma-Glutamyl Transferase (GGT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - LDH | Week 3
  - Hepatic workup: Lactate Dehydrogenase (LDH) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - ALP | Week 3
  - Hepatic workup: Alkaline Phosphatase (ALP) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - bilirubin | Week 3
  - Hepatic workup: Bilirubin (free/conjugated) concentration will be measured il micromoles/L
Intercycle report : Liver in Cohort 2 - AST | Week 3
  - Hepatic workup: Aspartate Aminotransferase (AST) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - ALT | Week 3
  - Hepatic workup: Alanine Aminotransferase (ALT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - GGT | Week 3
  - Hepatic workup: Gamma-Glutamyl Transferase (GGT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - LDH | Week 3
  - Hepatic workup: Lactate Dehydrogenase (LDH) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - ALP | Week 3
  - Hepatic workup: Alkaline Phosphatase (ALP) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - bilirubin | Week 3
  - Hepatic workup: bilirubin (free/conjugated) concentration will be measured in micromoles/L.
Intercycle report : Creatinine Phosphokinase in Cohort 1 | Week 3
  Creatine Phosphokinase will be measured in IU/L. usually between 60 and 400 IU/L
Intercycle report : Creatinine Phosphokinase in Cohort 2 | Week 3
  Creatine Phosphokinase will be measured in IU/L. usually between 60 and 400 IU/L
Intercycle report : Thyroid in Cohort 1 | Week 3
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report : Thyroid in Cohort 2 | Week 3
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report : Cortisol in Cohort 1 | Week 3
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report : Cortisol in Cohort 2 | Week 3
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report : C-reactive protein in Cohort 1 | Week 3
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report : C-reactive protein in Cohort 2 | Week 3
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report : Urine in Cohort 1 | Week 3
  Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows:
  (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report : Urine in Cohort 2 | Week 3
  Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows:
  (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report: N-BNP, troponin in Cohort 1 | Week 3
  Serum N-BNP and troponin concentrations will be measured. These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.
Intercycle report: N-BNP, troponin in Cohort 2 | Week 3
  Serum N-BNP and troponin concentrations will be measured.These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.
Intercycle report: Blood cells & platelets in Cohort 1 | Week 6
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report: Blood cells & Platelets in Cohort 2 | Week 6
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report: Electrolytes in Cohort 1 | Week 6
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report : Electrolytes in Cohort 2 | Week 6
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report : Liver in Cohort 1 - AST | Week 6
  Hepatic workup: Aspartate Aminotransferase (AST) concentration will be measured in IU/L..
Intercycle report : Liver in Cohort 1 - ALT | Week 6
  Hepatic workup: Aminotransferase (ALT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - GGT | Week 6
  Hepatic workup: Gamma-Glutamyl Transferase (GGT) concentrations will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - LDH | Week 6
  Hepatic workup: Lactate Dehydrogenase (LDH) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - ALP | Week 6
  Hepatic workup: Alkaline Phosphatase (ALP) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 1 - bilirubin | Week 6
  Hepatic workup: Bilirubin (free/conjugated) concentration will be measured in micromoles/L
Intercycle report : Liver in Cohort 2 - AST | Week 6
  - Hepatic workup: Aspartate Aminotransferase (AST) concentration will be measured.
Intercycle report : Liver in Cohort 2 - ALT | Week 6
  - Hepatic workup: Alanine Aminotransferase (ALT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - GGT | Week 6
  - Hepatic workup: Gamma-Glutamyl Transferase (GGT) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - LDH | Week 6
  - Hepatic workup: Lactate Dehydrogenase (LDH) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - ALP | Week 6
  - Hepatic workup: Alkaline Phosphatase (ALP) concentration will be measured in IU/L.
Intercycle report : Liver in Cohort 2 - bilirubin | Week 6
  - Hepatic workup: Bilirubin (free/conjugated) concentration will be measured in micromoles/L.
Intercycle report : Creatine Phosphokinase in Cohort 1 | Week 6
  - Creatine Phosphokinase will be measured in IU/L. Normal values are usually between 60 and 400 IU/L
Intercycle report : Creatine Phosphokinase in Cohort 2 | Week 6
  - Creatine Phosphokinase will be measured in IU/L. usually between 60 and 400 IU/L
Intercycle report : Thyroid in Cohort 1 | Week 6
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report : Thyroid in Cohort 2 | Week 6
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report : Cortisol in Cohort 1 | Week 6
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report : Cortisol in Cohort 2 | Week 6
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report : C-reactive protein in Cohort 1 | Week 6
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report : C-reactive protein in Cohort 2 | Week 6
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report : Urine in Cohort 1 | Week 6
  Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows:
  (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report : Urine in Cohort 2 | Week 6
  - Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows: (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report : N-BNP, troponin in Cohort 1 | Week 6
  Serum N-BNP and troponin concentrations will be measured.These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.
Intercycle report : N-BNP, troponin in Cohort 2 | Week 6
  Serum N-BNP and troponin concentrations will be measured.These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.
Intercycle report: Blood cells & Platelets in Cohort 1 | Week 9
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report: Blood cells & Platelets in Cohort 2 | Week 9
  The numbers of each type of blood cell and platelets will be measured per McL
Intercycle report: Electrolytes in Cohort 1 | Week 9
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report: Electrolytes in Cohort 2 | Week 9
  A basic metabolic panel will be run to measure Na, K, Cl and Protein levels.
Intercycle report: Liver in Cohort 1 | Week 9
  - Hepatic workup: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-Glutamyl Transferase (GGT), Lactate Dehydrogenase (LDH), Alkaline Phosphatase (ALP) and bilirubin (free/conjugated) concentrations will all be measured.
Intercycle report: Liver in Cohort 2 | Week 9
  - Hepatic workup: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-Glutamyl Transferase (GGT), Lactate Dehydrogenase (LDH), Alkaline Phosphatase (ALP) and bilirubin (free/conjugated) concentrations will all be measured.
Intercycle report: Creatine Phosphokinase in Cohort 1 | Week 9
  Creatine Phosphokinase Creatine Phosphokinase will be measured in IU/L. usually between 60 and 400 IU/L
Intercycle report: Creatine Phosphokinase in Cohort 2 | Week 9
  Creatine Phosphokinase will be measured in IU/L. usually between 60 and 400 IU/L
Intercycle report: Thyroid in Cohort 1 | Week 9
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report: Thyroid in Cohort 2 | Week 9
  A thyroid stimulating test (total T4 test) will be made to measure the thyroxine concentration in the patient's blood.
Intercycle report: Cortisol in Cohort 1 | Week 9
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report: Cortisol in Cohort 2 | Week 9
  Cortisol (serum) levels will be measured at 8 a.m. only (i.e. one cycle out of two) to check whether the adrenal glands are functioning correctly. Normal levels for adults in the morning are :
  5-25 mcg/dL (138-690 nmol/L) or 5-23 mcg/dL (138-635 nmol/L) for elderly patients.
Intercycle report: C-reactive protein in Cohort 1 | Week 9
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report: C-reactive protein in Cohort 2 | Week 9
  C-reactive protein will be measured in mg/L. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L).
Intercycle report : Urine in Cohort 1 | Week 9
  Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows:
  (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report: Urine in Cohort 2 | Week 9
  Urinary balance: via a cytobacteriological examination, the protein/creatinine ratio will be calculated as follows:
  (Urine protein(g/L) X 1000)/Urine creatinine(mmol/L)
Intercycle report: N-BNP, troponin in Cohort 1 | Week 9
  Serum N-BNP and troponin concentrations will be measured. These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.
Intercycle report: N-BNP, troponin in Cohort 2 | Week 9
  Serum N-BNP and troponin concentrations will be measured. These are biomarkers of heart failure. N-BNP is measured in pg/mL and troponin is measured in ng/mL.

OTHER OUTCOMES:
Tumor staging in Cohort 1 | Just before surgery at weeks 14 to 18
  Via computed tomographic urography, tumor classification will be performed using the 2017 TNM classification for upper urothelial tract carcinomas. High-risk UTUC is defined by risk stratification following EAU guidelines. Endoluminal filling defects surrounded by opacified urine will be considered as non-infiltrative lesions corresponding to Stage T1. Focal thickening of the urethral wall or renal pelvis = Stage T2. Fat infiltration in front of the parietal thickening or infiltration of kidney tissue = Stage T3.
Tumor staging in Cohort 2 | Just before surgery at weeks 14 to 18
  Via computed tomographic urography, tumor classification will be performed using the 2017 TNM classification for upper urothelial tract carcinomas. High-risk UTUC is defined by risk stratification following EAU guidelines. Endoluminal filling defects surrounded by opacified urine will be considered as non-infiltrative lesions corresponding to Stage T1. Focal thickening of the urethral wall or renal pelvis = Stage T2. Fat infiltration in front of the parietal thickening or infiltration of kidney tissue = Stage T3.
Results of biopsy on tissue specimens after surgery in Cohort 1 | After surgery at weeks 14 to 18
  After surgery, paraffin-embedded tissues and tissues frozen to -80° obtained during surgery will be evaluated by Ventana 623 assay. The PD-L1 status of both tumor cells and immune cells will be recorded.
Results of biopsy on tissue specimens after surgery in Cohort 2 | After surgery at weeks 14 to 18
  After surgery, paraffin-embedded tissues and tissues frozen to -80° obtained during surgery will be evaluated by Ventana 623 assay. The PD-L1 status of both tumor cells and immune cells will be recorded.
Overall survival in Cohort 1 | Approximately two years after surgery
  The overall survival rate of patients in Cohort 1 will be noted following a phone-call to the patient's home. If the patient has died, information regarding the cause of death will be sought from the INSERM's Cepi-DC file (where all records of deceased patients are kept).
Overall survival in Cohort 2 | Approximately two years after surgery
  The overall survival rate of patients in Cohort 2 will be noted following a phone-call to the patient's home.If the patient has died, information regarding the cause of death will be sought from the INSERM's Cepi-DC file (where all records of deceased patients are kept).
Bladder recurrence in Cohort 1 | Approximately two years after surgery
  A phone-call to the patient's home will be made and any bladder recurrence will be noted.
Bladder recurrence in Cohort 2 | Approximately two years after surgery
  A phone-call to the patient's home will be made and any bladder recurrence will be noted.
Dissemination in Cohort 1 | Approximately two years after surgery
  A phone-call to the patient's home will be made and any tumor dissemination will be noted.
Dissemination in Cohort 2 | Approximately two years after surgery
  A phone-call to the patient's home will be made and any tumor dissemination will be noted.

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Hôpital Bichat-Claude Bernard, Paris, Paris Cx 20
  - Institut Paoli Calmette, Marseille
  - Hôpital Saint Louis, Paris
  - Hôpital Pitié Salpétrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Hôpital Foch, Suresnes
  - Iuct Oncopole, Toulouse

REFERENCES:
- [Derived] Houede N, Chevallier T, Audenet F, Thibault C, Neuzillet Y, Abraham C, Masson-Lecomte A, Gauthier H, Gravis G, Pignot G, Tartas S, Ruffion A, Pouessel D, Roumiguie M, Laguerre B, Bensalah K, Xylinas E, Jaffrelot L, Droupy S, Luquiens G, Roupret M. Safety and Efficacy of Neoadjuvant Durvalumab Plus Gemcitabine/Cisplatin or Carboplatin in Patients With Operable High-Risk Upper Tract Urothelial Carcinoma: The iNDUCT-GETUG V08 Trial. J Clin Oncol. 2025 May;43(13):1578-1586. doi: 10.1200/JCO-25-00179. Epub 2025 Feb 14. PMID 39951246
- [Derived] Calleris G, Roupret M, Seisen T, Bendjeddou L, Chevallier T, Masson-Lecomte A, Thibault C, Neuzillet Y, Audenet F, Xylinas E, Houede N. Design and rationale of a single-arm phase II study of neoadjuvant Durvalumab and Gemcitabine associated with Cisplatin or Carboplatin for upper urinary tract urothelial cancer: the iNDUCT trial (NCT04617756). World J Urol. 2023 Dec;41(12):3413-3420. doi: 10.1007/s00345-023-04596-5. Epub 2023 Sep 12. PMID 37698632